CLINICAL TRIAL: NCT03604211
Title: Predictive Factors for the Benefit of Stereotactic Body Radiotherapy for Oligometastatic Lymph Node Recurrence in Prostate Cancer: a Single Institution Experience
Brief Title: SBRT for Oligometastatic Lymph Node Recurrence in Prostate Cancer: a Single Institution Experience
Status: Completed | Type: Observational
Sponsor: Kantonsspital Graubuenden (Other)
Collaborators: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: KGraubuenden
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer Recurrent; Prostate Cancer; Lymph Node Metastases
MeSH Terms: conditions — Prostatic Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Cyberknife Radiation Therapy — Stereotactic Radiotherapy of lymphnode recurrence after prostatectomy +/- salvage radiotherapy

SUMMARY:
Single-institution retrospective analysis for predictive factors of prostate cancer patients presenting with isolated or limited lymph node (LN) recurrence (1-3 lesions) on F-Ccholine PET-CT (CholPET) treated with SBRT between January 2010 and July 2015.

DETAILED DESCRIPTION:
Single-institution retrospective analysis of consecutive prostate cancer patients after definitive primary treatment, without local recurrence, presenting with isolated or limited lymph node (LN) recurrence (1-3 lesions) on F-Ccholine PET-CT (CholPET) treated with SBRT between January 2010 and July 2015.

Endpoints of interest are biochemical response rate (defined as a reduction by at least 10% of the initial PSA value), time to biochemical recurrence (TBR) (defined as the time interval from SBRT until second PSA rise), and time interval between SBRT and ADT start. Univariate analysis is used to identify prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven diagnosis of prostate cancer
* Radical prostatectomy (± salvage radiotherapy)
* PSA relapse (defined by two consecutive rising PSA values >0.2 ug/l)
* one to three lymphnodes positive on Choline-PET
* no recurrence in prostatic bed on Choline-PET
* WHO performance status of 0-1
* no previous chemotherapy or ADT for prostate cancer.

Exclusion Criteria:

* primary treatment for prostate cancer by RT or brachytherapy
* bone (M1b) metastases
* visceral (M1c) metastases
* any symptomatic nodal lesion

Ages: 18 Years to 85 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: single-Institution cohort of male patients 18-85 years of age, with recurrent prostate cancer after radical prostatectomy in 1-3 lymphnodes, prospectively registered in a local institutional database
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
time to biochemical recurrence | 18 months
  time interval from SBRT until second PSA rise

SECONDARY OUTCOMES:
biochemical response rate | 18 months
  reduction by at least 10% of the initial PSA value
time interval between SBRT and ADT start | 18 months
  time interval between SBRT and ADT start

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Zwahlen, MD, Study Director — Kantonsspital Graubuenden
Locations (1):
- Juergen Curschmann, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No